CLINICAL TRIAL: NCT07049926
Title: A Phase 1b/2 Study of Immune and Targeted Combination Therapies in Participants With RCC (KEYMAKER-U03): Substudy 03C in Participants With Recurrent Disease During or After Anti-PD-(L)1 Adjuvant Therapy
Brief Title: Substudy 03C: A Study of Combination Therapies in Participants With Renal Cell Carcinoma With Recurrent Disease During or After Anti-PD-(L)1 Therapy (MK-3475-03C/KEYMAKER-U03)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3475-03C; MK-3475-03C (Other: MSD); 2024-516437-12-00 (Registry Identifier: EU CT); U1111-1310-6076 (Registry Identifier: UTN); KEYMAKER-U03 (Other: MSD)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma
Keywords: Vascular Endothelial Growth Factor Receptor-Tyrosine Kinase Inhibitor (VEGFR-TKI); Hypoxia-Inducible Factor-2α (HIF-2α)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — belzutifan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zanzalintinib at Dose Level 1 or 2 + Belzutifan (Experimental): Participants will be allocated to receive zanzalintinib at dose level 1 or 2 + belzutifan daily until progressive disease or discontinuation
  Interventions: Drug: Belzutifan; Drug: Zanzalintinib
- Belzutifan (Experimental): Participants will receive belzutifan daily until progressive disease or discontinuation
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Oral Tablet
  Other Names: WELIREG®; MK-6482; PT2977
Drug: Zanzalintinib — Oral Tablet
  Other Names: XL092
  Arms: Zanzalintinib at Dose Level 1 or 2 + Belzutifan

SUMMARY:
Substudy 03C is part of a larger research study that is testing experimental treatments for renal cell carcinoma (RCC). The larger study is the umbrella study (U03).

The goal of substudy 03C is to evaluate the safety and efficacy of experimental combinations of investigational agents in participants with clear cell renal cell carcinoma (ccRCC) who have recurrent disease during or after anti-programmed cell death 1/programmed cell death ligand 1 (PD-[L]1) adjuvant therapy.

This substudy will have two phases: a safety lead-in phase and an efficacy phase. The safety lead-in phase will be used to demonstrate a tolerable safety profile for the combination of investigational agents. There will be no hypothesis testing in this study

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Has a histologically confirmed diagnosis of unresectable locally advanced/metastatic renal cell carcinoma (RCC) with clear cell component
* Has received no other prior systemic therapy for treatment of advanced/metastatic clear cell renal cell carcinoma (ccRCC) except for adjuvant programmed cell death ligand 1 (PD-(L)1) therapy
* Has disease recurrence during adjuvant anti- PD-(L)1 therapy or ≤24 months following the last dose of adjuvant anti-PD-(L)1 therapy
* Is able to swallow oral medication
* Submits an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Participants receiving bone resorptive therapy (must have therapy initiated at least 2 weeks before allocation/randomization)
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤140/90 mm Hg with no change in antihypertensive medications within 1 week before allocation/randomization
* Has adequate organ function

The main exclusion criteria include but are not limited to the following:

* Has clinically significant hematuria, hematemesis, or hemoptysis of (>2.5 mL) of red blood, or other history of significant bleeding
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention
* Has deep vein thrombosis within 3 months before allocation/randomization unless stable, asymptomatic, and treated with therapeutic anticoagulation for at least 4 weeks before allocation/randomization
* Has history of idiopathic pulmonary fibrosis, organizing pneumonia, or evidence of active pneumonitis
* Has serious wound, ulcer or bone fracture or has had major surgery within 8 weeks before first dose of study intervention
* Has symptomatic pleural effusion (for example cough, dyspnea, pleuritic chest pain), ascites, or pericardial fluid requiring drainage in the last 4 weeks before allocation/randomization
* Has gastrointestinal (GI) disorders, including those associated with a high risk of perforation or fistula formation
* Has malabsorption due to prior GI surgery or GI disease
* Has moderate to severe hepatic impairment
* Has received colony-stimulating factors within 28 days prior to intervention allocation/randomization
* Has received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Is currently receiving strong inhibitors of cytochrome P450 3A4 (CYP3A4) that cannot be discontinued for the duration of the study
* Has received a live or live attenuated vaccine within 30 days before the first dose of study intervention
* Is currently receiving anticoagulants or platelet inhibitors that cannot be discontinued for the duration of the study
* Have been previously allocated/randomized to study intervention in any sub study of protocol MK-3475-U03
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has an active infection requiring systemic therapy
* Has history of human immunodeficiency virus (HIV) infection
* Has hepatitis B or hepatitis C virus infection

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2031-10-26 (Estimated); Study Completion 2031-10-26 (Estimated)

PRIMARY OUTCOMES:
Safety Lead In Phase: Number of participants who experience one or more dose-limiting toxicities (DLTs) | Up to approximately 21 days
  DLTs are defined as any of a pre-specified list of toxicities if assessed by the investigator to be possibly, probably, or definitely related to study treatment administration, excluding toxicities clearly not related to the drug, such as disease progression, environmental factors, unrelated trauma, etc.
Safety Lead In Phase: Number of participants who experience one or more adverse events (AEs) | Up to approximately 74 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Safety Lead In Phase: Number of participants who discontinue study treatment due to an AE | Up to approximately 74 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Efficacy Phase: Number of participants who experience one or more DLTs | Up to approximately 21 days
  DLTs are defined as any of a pre-specified list of toxicities if assessed by the investigator to be possibly, probably, or definitely related to study treatment administration, excluding toxicities clearly not related to the drug, such as disease progression, environmental factors, unrelated trauma, etc.
Efficacy Phase: Number of participants who experience one or more AEs | Up to approximately 74 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Efficacy Phase: Number of participants who discontinue study treatment due to an AE | Up to approximately 74 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Efficacy Phase: Objective Response Rate (ORR) | Up to approximately 74 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Efficacy Phase: Duration of response (DOR) | Up to approximately 74 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Efficacy Phase: Progression-free survival (PFS) | Up to approximately 74 months
  PFS is defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Efficacy Phase: Overall survival (OS) | Up to approximately 74 months
  OS is defined as time from first dose of study treatment to death due to any cause.
Efficacy Phase: Clinical benefit rate (CBR) | Up to approximately 74 months
  CBR is defined as the percentage of participants who have achieved stable disease (SD: Neither sufficient shrinkage to qualify for PR [at least a 30% decrease in the sum of diameters of target lesions] nor sufficient increase to qualify for PD) of ≥6 months or confirmed CR (disappearance of all target lesions) or PR per RECIST 1.1. PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The CBR as assessed by BICR will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (23):
- United States (5):
  - UCSF Medical Center at Mission Bay ( Site 5008), San Francisco, California
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 5026), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center ( Site 5016), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 5002), New York, New York
  - Duke Cancer Institute ( Site 5015), Durham, North Carolina
- France (4):
  - Institut Claudius Regaud ( Site 5200), Toulouse, Haute-Garonne
  - Centre Eugene Marquis ( Site 5205), Rennes, Ille-et-Vilaine
  - Institut De Cancerologie De Lorraine ( Site 5204), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Gustave Roussy ( Site 5202), Villejuif, Île-de-France Region
- Israel (4):
  - Rambam Health Care Campus ( Site 5500), Haifa
  - Rabin Medical Center ( Site 5502), Petah Tikva
  - Sheba Medical Center ( Site 5501), Ramat Gan
  - Sourasky Medical Center ( Site 5503), Tel Aviv
- Poland (2):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 6201), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 6202), Gdansk, Pomeranian Voivodeship
- South Korea (3):
  - Severance Hospital ( Site 5802), Seoul
  - Asan Medical Center ( Site 5800), Seoul
  - Samsung Medical Center ( Site 5801), Seoul
- Spain (2):
  - Hospital Universitario Ramon y Cajal ( Site 5301), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron ( Site 5300), Barcelona
- United Kingdom (3):
  - Western General Hospital ( Site 5402), Edinburgh, Edinburgh, City of
  - St Bartholomew's Hospital ( Site 5401), London, London, City of
  - The Christie NHS Foundation Trust ( Site 5400), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/